CLINICAL TRIAL: NCT03892044
Title: A Phase I Study of Duvelisib in Combination With Nivolumab for Patients With Richter's Syndrome and Transformed Follicular Lymphoma
Brief Title: Duvelisib and Nivolumab in Treating Patients With Richter Syndrome or Transformed Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Bond, MD (Other)
Responsible Party: Sponsor-Investigator, David Bond, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18173; NCI-2019-01028 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Richter Syndrome; Small Lymphocytic Lymphoma; Transformed Chronic Lymphocytic Leukemia to Diffuse Large B-Cell Lymphoma; Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Transformed Small Lymphocytic Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — duvelisib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (duvelisib, nivolumab) (Experimental): Patients receive duvelisib PO BID on days 1-28 and nivolumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Duvelisib; Biological: Nivolumab

INTERVENTIONS:
Drug: Duvelisib — Given PO
  Other Names: 8-Chloro-2-phenyl-3-((1S)-1-(7H-purin-6-ylamino)ethyl)isoquinolin-1(2H)-one; INK-1197; IPI-145
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase I trial studies the side effects and best dose of duvelisib when given together with nivolumab in treating patients with Richter syndrome or transformed follicular lymphoma. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving duvelisib and nivolumab may work better in treating patients with Richter syndrome or transformed follicular lymphoma compared to giving duvelisib or nivolumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) of duvelisib in combination with nivolumab for patients with Richter?s syndrome or transformed follicular lymphoma.

SECONDARY OBJECTIVES:

I. To assess preliminary efficacy of duvelisib in combination with nivolumab in Richter?s syndrome and transformed follicular lymphoma (overall response rate, progression free survival, overall survival).

II. To determine the toxicity profile of duvelisib in combination with nivolumab.

EXPLORATORY OBJECTIVES:

I. To correlate response to duvelisib in combination with nivolumab with cytogenetic/fluorescence in-situ hybridization (FISH) abnormalities of the chronic lymphocytic leukemia (CLL) and lymphoma compartments (for patients with Richter?s syndrome) at baseline.

II. To correlate response to duvelisib in combination with nivolumab with baseline deoxyribonucleic acid (DNA) mutation of CLL and lymphoma as assessed in tumor samples and cell free DNA.

III. To determine changes in T, B, and natural killer (NK) cell number and function during duvelisib plus nivolumab therapy.

OUTLINE: This is a dose-escalation study of duvelisib.

Patients receive duvelisib orally (PO) twice daily (BID) on days 1-28 and nivolumab intravenously (IV) over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL or small lymphocytic lymphoma (SLL) meeting International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria AND biopsy proven transformation to diffuse large B cell lymphoma (DLBCL), clinically consistent with Richter?s syndrome (RS) OR histologically diagnosed relapsed or refractory DLBCL including transformed follicular lymphoma (tFL) ineligible for or refractory to platinum containing salvage therapy for the dose escalation portion of the study. For the dose expansion phase only patients with CLL with transformation to DLBCL or tFL will be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 500/uL
* Platelet count >= 30,000/uL (unless due to bone marrow involvement)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 ULN
* Total bilirubin =< 1.5 ULN (unless due to liver involvement, hemolysis, or Gilbert?s disease)
* Creatinine clearance >= 40 mL/min (Cockcroft-Gault estimated)
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study
* Patients must sign an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Documented infection with human immunodeficiency virus (HIV) or chronic, active hepatitis B or C infection
* Any chemotherapy or monoclonal antibodies within 14 days or kinase inhibitors (except BTKi) within 5 half-lives before cycle 1, day 1 (C1D1). BTK inhibitors may be continued until 2 days prior to C1D1. Steroids are allowed for palliation of symptoms due to lymphoma
* Toxicity from previous therapy which has not resolved to grade 1 (or patient?s previous baseline)
* Other active malignancies except those treated with curative intent with no active disease at the time of study entry or those felt to be at low risk of progression or recurrence over the next 2 years (such as low risk prostate cancer on active surveillance)
* New York Heart Association (NYHA) class III/IV heart disease or other significant medical condition or organ system dysfunction which could compromise the subject?s safety or put the study outcomes at undue risk
* Uncontrolled systemic infection
* Unable to swallow capsules or significant malabsorption syndrome, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction at the time of screening
* Patients who are pregnant or breastfeeding
* Patients with known central nervous system (CNS) involvement by CLL or lymphoma
* Patients who have underwent autologous or allogeneic stem cell transplant =< 4 weeks prior to C1D1 or have active graft-versus-host disease are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of duvelisib | Up to 28 days
  The MTD is defined as the highest dose level where at most one patient out of six experiences dose-limiting toxicities.

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years
  Will be defined as the proportion of patients achieving a complete or partial response; any eligible patient who begins treatment with the combination regimen will be included in the denominator. Will be calculated with a 95% binomial confidence interval.
Progression-free survival (PFS) | From cycle 1, day 1 to date of progression or death, assessed up to 3 years
  The method of Kaplan Meier will be used to estimate PFS.
Overall survival (OS) | From cycle 1, day 1 to date of progression or death, assessed up to 3 years
  The method of Kaplan Meier will be used to estimate OS.

OTHER OUTCOMES:
Response to duvelisib in combination with nivolumab | Baseline
  Will be correlated with cytogenetic/fluorescence in-situ hybridization abnormalities of the chronic lymphocytic leukemia (CLL) and lymphoma compartments (for patients with Richter syndrome). The chi-squared test and logistic regression will be utilized to evaluate the association.
Response to duvelisib in combination with nivolumab | Baseline
  Will be correlated with deoxyribonucleic acid (DNA) mutation of CLL and lymphoma and assessed in tumor samples and cell free DNA. The chi-squared test and logistic regression will be utilized to evaluate the association.
Changes in T, B, and NK cell number and function | Up to 3 years
  Will be summarized using graphical method in a descriptive manner and tested using nonparametric Wilcoxon signed-rank test due to small sample size.

CONTACTS AND LOCATIONS:
Overall Officials: David Bond, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannello A, Vitale N, Coma S, Arruga F, Chadburn A, Di Napoli A, Laudanna C, Allan JN, Furman RR, Pachter JA, Deaglio S, Vaisitti T. Synergistic efficacy of the dual PI3K-delta/gamma inhibitor duvelisib with the Bcl-2 inhibitor venetoclax in Richter syndrome PDX models. Blood. 2021 Jun 17;137(24):3378-3389. doi: 10.1182/blood.2020010187. PMID 33786583
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03892044/ICF_000.pdf